CLINICAL TRIAL: NCT00716872
Title: Evaluating Internet-Based Interventions for Insomnia in Cancer Patients
Brief Title: Improving the Sleep of Cancer Patients Using an Internet-Based Program
Acronym: SHUTi-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Lee Ritterband, Ph.D., University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13685
Record Dates: First submitted 2008-06-18; First posted 2008-07-16 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Cancer; Insomnia
Keywords: cancer; sleep; insomnia; Internet; SHUTi
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ImmedSHUTi/ImmedHyp (Experimental): In the first part of the trial, participants are assigned to the Immediate SHUTi group; that is, they receive access to the SHUTi program right away. In the second part of the trial (3 months later), participants are assigned to the Immediate Hypnosis group; that is, they receive access to the Hypnosis recordings right away.
  Interventions: Behavioral: Sleep Healthy Using the Internet (SHUTi); Behavioral: Hypnosis recordings
- ImmedSHUTi/DelayHyp (Experimental): In the first part of the trial, participants are assigned to the Immediate SHUTi group; that is, they receive access to the SHUTi program right away. In the second part of the trial (3 months later), participants are assigned to the Delayed Hypnosis group; that is, they receive access to the Hypnosis recordings at the end of the study.
  Interventions: Behavioral: Sleep Healthy Using the Internet (SHUTi)
- DelaySHUTi/ImmedHyp (Experimental): In the first part of the trial, participants are assigned to the Delayed SHUTi group; that is, they receive access to the SHUTi program at the end of the study. In the second part of the trial (3 months later), participants are assigned to the Immediate Hypnosis group; that is, they receive access to the Hypnosis recordings right away.
  Interventions: Behavioral: Hypnosis recordings
- DelaySHUTi/DelayHyp (No Intervention): In the first part of the trial, participants are assigned to the Delayed SHUTi group; that is, they receive access to the SHUTi program at the end of the study. In the second part of the trial (3 months later), participants are assigned to the Delayed Hypnosis group; that is, they receive access to the Hypnosis recordings at the end of the study.

INTERVENTIONS:
Behavioral: Sleep Healthy Using the Internet (SHUTi) — SHUTi is an Internet program based on cognitive-behavioral therapy for insomnia (CBT-I). Users complete daily online sleep diaries in addition to receiving weekly access to six interactive "Cores" of information. As they progress through the program, users receive tailored instructions for how to improve their sleep.
  Arms: ImmedSHUTi/DelayHyp; ImmedSHUTi/ImmedHyp
Behavioral: Hypnosis recordings — Subjects listen to self-hypnosis recordings designed to improve their disturbed sleep.
  Arms: DelaySHUTi/ImmedHyp; ImmedSHUTi/ImmedHyp

SUMMARY:
The purpose of this study is to determine whether an Internet-based program, Sleep Healthy Using the Internet (SHUTi, or "Shut-Eye"), can help to improve the sleep of people who are in remission from cancer and experiencing symptoms of insomnia.

DETAILED DESCRIPTION:
The purpose of this study is to test the feasibility of using an Internet program to improve the sleep of cancer patients with insomnia. Participants will receive access to the Internet program (called SHUTi, or "Shut-Eye") as well as to self-hypnosis recordings designed to improve sleep. SHUTi provides an online, tailored educational program to individuals who are experiencing sleep difficulties, including those having difficulty falling asleep, waking in the middle of the night, and waking too early in the morning.

ELIGIBILITY:
Inclusion Criteria:

* Age = At least 21 years old
* Regular access to the Internet, including e-mail
* Cancer patient

  * Any type of cancer (EXCEPT non-melanoma skin cancer)
  * In remission from any stage of cancer (active treatment completed at least one month prior to enrollment)
* Insomnia diagnosis (combined from DSM-IV and ICSD):

  * Subjective complaints of poor sleep for at least 6 months
  * Sleep difficulties ≥3 nights/week
* Difficulty falling asleep (≥30 minutes to fall asleep) OR
* Difficulty staying asleep (≥30 minutes awake in the middle of the night)

  * ≤6.5 hours sleep/night
  * Poor sleep causes marked distress or significant impairment in daytime functioning (e.g. fatigue, performance deficits, mood disturbance)
* Participant feels that the insomnia was caused/aggravated by cancer or cancer treatment

Exclusion Criteria:

* Having a sleep disorder other than insomnia (e.g. sleep apnea, RLS, narcolepsy, parasomnias)
* Having a medical condition other than cancer that causes insomnia
* Experiencing a psychiatric disturbance (major depression, psychosis)
* Experiencing substance abuse
* Currently undergoing psychotherapy or counseling
* Changing sleep/anxiety/depression medication within the past month
* Having an "unusual" sleep pattern

  * Normal bedtime is after 2am OR
  * Normal wake time is after 9am
* Working as a shift worker (that is, having a schedule that requires working through the night)
* Participants reports that she is pregnant or intending to get pregnant in the next 4 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | prior to intervention, after SHUTi use, after Hypnosis use
Sleep Diary: Sleep Efficiency | prior to intervention, after SHUTi use, after Hypnosis use
Sleep Diary: Total Sleep Time | prior to intervention, after SHUTi use, after Hypnosis use

SECONDARY OUTCOMES:
Sleep Diary: Sleep Onset Latency (SOL) | prior to intervention, after SHUTi use, after Hypnosis use
Sleep Diary: Wake After Sleep Onset (WASO) | prior to intervention, after SHUTi use, after Hypnosis use
Sleep Diary: Number of Nighttime Awakenings | prior to intervention, after SHUTi use, after Hypnosis use
Hospital Depression and Anxiety Scale | prior to intervention, after SHUTi use, after Hypnosis use
Pain scale | prior to intervention, after SHUTi use, after Hypnosis use
Multidimensional Fatigue Symptom Inventory | prior to intervention, after SHUTi use, after Hypnosis use
Quality of Life (SF-12 Health Survey) | prior to intervention, after SHUTi use, after Hypnosis use
Hot flashes | prior to intervention, after SHUTi use, after Hypnosis use

CONTACTS AND LOCATIONS:
Overall Officials: Lee M Ritterband, Ph.D., Principal Investigator — University of Virginia; Lora D Baum, Ph.D., Principal Investigator — University of Virginia; Elaine T Bailey, Ph.D., Study Director — University of Virginia
Locations (1):
- University of Virginia Department of Psychiatry & Neurobehavioral Sciences, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Savard J, Simard S, Ivers H, Morin CM. Randomized study on the efficacy of cognitive-behavioral therapy for insomnia secondary to breast cancer, part I: Sleep and psychological effects. J Clin Oncol. 2005 Sep 1;23(25):6083-96. doi: 10.1200/JCO.2005.09.548. PMID 16135475